CLINICAL TRIAL: NCT03046186
Title: Effect of Gastric Sleeve Operation on Absorption and Metabolism of Glucose and Protein as Well as Gut-hormonal Response - A Comparison With Roux-en-Y Gastric Bypass
Brief Title: Physiological Effects of Gastric Sleeve Operation
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, MD, Hvidovre University Hospital
Other Study IDs: MS-SGRYGB-15
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Obesity, Morbid; Bariatric Surgery
Keywords: Gastric sleeve; Gastric bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine samples during mixed meal test with double tracer tecnique using iv tracers ([D2] Phenylalanine, [ring-D4]Tyrosine, [6,6-2H2]Glucose, [1,1,2,3,3-2H5]Glycerol, [15N2]Urea and labelled oral tracers ([U13C6]glucose, intrinsically [ring-D5]Phenylalanine).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastric sleeve operated subjects: 12 patients who have undergone gastric sleeve operation >12 month prior to inclution.
  Interventions: Diagnostic Test: Mixed meal test with double tracer technique
- Control Subjects: 12 Healthy un-operated control subjects matched to the gastric sleeve group in a one to one manner with respect to BMI, sex and age
  Interventions: Diagnostic Test: Mixed meal test with double tracer technique
- Gastric bypass operated subjects: 12 patients, who have undergone Roux-en-Y gastric bypass >12 month prior to inclution, matched to the gastric sleeve group in a one to one manner with respect to pre-operative BMI, post-operative BMI, sex and age.
  Interventions: Diagnostic Test: Mixed meal test with double tracer technique

INTERVENTIONS:
Diagnostic Test: Mixed meal test with double tracer technique

SUMMARY:
After gastric sleeve patients undergo a substantial weight loss, but the physiological mechanisms behind the weight loss is not fully elucidated. Studies suggest that gut-hormone secretion is altered comparable to what is also seen after Roux-en-Y gastric bypass, however to which extent is not fully established and furthermore, the mechanisms behind an altered secretion are unclear. The purpose of this study is to investigate absorption and postprandial metabolism of glucose and protein in addition to gut hormonal responses after gastric sleeve compared with a group of un-operated subjects machted on sex, age and BMI. Furter, a group of Roux-en-Y gastric bypass operated patients matched on pre-operative BMI, current BMI, sex and age will be included for comparison.

ELIGIBILITY:
SG ang RYGB group:

Inclusion Criteria:

* Uncomplicated RYGB or SG > 12 month prior to inclusion
* Weight stable (+/- 3 month the last month)
* Written informed consent

Exclusion Criteria:

* Diabetes (HbA1c>48 or Fasting plasma-glucose>6.1 mM)
* Pregnancy and/or breastfeeding
* Inadequately treated thyroid disease
* Serious heart or respiratory illness
* Haemoglobin < 6,5 mM.

Un-operated control group:

Inclusion Criteria:

* Written informed consent

Exclusion Criteria:

* Prior RYGB, SG or complicated upper gastrointestinal surgery
* Diabetes (HbA1c>48 or Fasting plasma-glucose>6.1 mM)
* Pregnancy and/or breastfeeding
* Inadequately treated thyroid disease
* Serious heart or respiratory illness
* Haemoglobin < 6,5 mM.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients, who have undergone Roux-en-Y gastric bypass OR gastric sleeve operation > 12 month prior to inclusion.
  Matched un-operated control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Glucose absorption | 0 - 360 minutes
  Between groups difference in peak Rate of appearance (Ra) of oral glucose tracer SG vs. CON
Protein absorption | 0 - 360 minutes
  Between groups difference in peak Ra of oral aminoacid tracer SG vs. CON

SECONDARY OUTCOMES:
Glucose absorption | 0 - 360 minutes
  Between group difference in peak Ra of oral glucose comparing SG vs. RYGB
Protein absorption | 0 - 360 minutes
  Between groups differences in peak Ra of oral aminoacid tracer comparing SG vs. RYGB
Glucose kinetics | 0 - 360 minutes
  Between groups differences in AUC Ra of oral glucose tracer
Protein kinetics | 0 - 360 minutes
  Between groups differences in AUC Ra of oral aminoacid tracer
Insulin secretion | 0 - 240 minutes
  Between groups differences in iAUC of serum insulin and C-peptide
Glucagon-like Peptide 1 (GLP-1) secretion | 0 - 240 minutes
  Between groups differences in iAUC of plasma concentration of GLP-1
Glucose-dependent Insulinotropic Peptide (GIP) | 0 - 240 minutes
  Between groups differences in iAUC of plasma concentration of GIP
Ghrelin secretion | 0 - 240 minutes
  Between groups differences in iAUC of plasma concentration of ghrelin
Glucagon secretion | 0-240 minutes
  Between groups differences in iAUC of plasma cncentration of glucagon
Peptide YY | 0-240 minutes
  Between groups differences in iAUC of plasma concentration of PYY
Endogenous glucose production | -120 - 360 minutes
  Calculated via double tracer tecnique both in the fasting and post prandial state.
Lipolysis | -120 - 360
  Between groups differences in Rate of Disappearance of glycerol tracer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Please Select, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svane MS, Bojsen-Moller KN, Martinussen C, Dirksen C, Madsen JL, Reitelseder S, Holm L, Rehfeld JF, Kristiansen VB, van Hall G, Holst JJ, Madsbad S. Postprandial Nutrient Handling and Gastrointestinal Hormone Secretion After Roux-en-Y Gastric Bypass vs Sleeve Gastrectomy. Gastroenterology. 2019 May;156(6):1627-1641.e1. doi: 10.1053/j.gastro.2019.01.262. Epub 2019 Feb 8. PMID 30742833